CLINICAL TRIAL: NCT06835985
Title: sIRB: Social Media Intervention for Online Victimized Youth
Brief Title: Social Media Intervention for Online Victimized Youth
Acronym: SMILEY
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Children's Hospital of Philadelphia (Other); University of Oregon (Other)
Responsible Party: Principal Investigator, César Escobar-Viera, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22040038; P50MH115838 (NIH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Depression; Suicidal Ideation
Keywords: online victimization; chatbot; social media intervention
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Participants will only be assigned to one of two interventions to compare SMILEY + brief psychoeducation (intervention) vs. brief psychoeducation (control).
Who Masked: Outcomes Assessor
Masking Description: Participants will know which of the two interventions they are being assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMILEY + Brief Psychoeducation (Experimental): SMILEY (Social Media Intervention for Online Victimized Youth): A self-paced HIPAA-compliant chatbot intervention administered through Facebook Messenger that delivers psychoeducational and coping skills content to improve social media self-efficacy and distress tolerance among Black, SGM and other minority youth with moderate to severe depression who experience online victimization.
  Interventions: Other: Chatbot Intervention; Other: Brief Psychoeducation
- Brief Psychoeducation (Active Comparator): Research clinician will deliver psychoeducation for youth and caregivers supported by web-based resources. Content will introduce basic concepts of social media self-efficacy (screen time guidance, technological coping skills, and encouragement of positive online interactions) and guidance on how to respond to and cope with online victimization.
  Interventions: Other: Brief Psychoeducation

INTERVENTIONS:
Other: Chatbot Intervention — Participants screened for suicidality during the ETUDES Center Primary Care Study and who disclose experiencing online victimization will be onboarded by a research clinician on how to use SMILEY, the web-based intervention that delivers psychoeducation, basic concepts of social media self-efficiency, and guidance on how to respond to and cope with online victimization. The chatbot and/or research clinician will send out periodic reminders to users to remind them to engage with the chatbot over four weeks. Technical troubleshooting concerns will be carried out by research clinician and chatbot developer team.
  Other Names: SMILEY
  Arms: SMILEY + Brief Psychoeducation
Other: Brief Psychoeducation — When youth onboard the study, a research clinician will deliver psychoeducation for youth and caregivers supported by web-based resources. Content will introduce basic concepts of social media self-efficacy (screen time guidance, technological coping skills, and encouragement of positive online interactions) and guidance on how to respond to and cope with online victimization.

SUMMARY:
This feasibility pilot trial seeks to examine the feasibility and target engagement of a coping skills and psychoeducational intervention delivered via an automated conversational chatbot named SMILEY in reducing frequency and stress associated with online victimization among marginalized youth, including those who are Black, Hispanic, and LGBTQ+, and experiencing depression and online victimization.

The primary inquiry of this study is whether SMILEY can enhance the safety and decrease stress levels in online environments for marginalized youth coping with depression and online victimization.

Participants will engage with materials, including interactive web resources, to learn safe social media practices and provide coping skills for experiencing online victimization. These materials will cover topics such as managing online time, addressing negative comments, and fostering positive connections.

Participants will interact with SMILEY at their own pace over 4 weeks. This interaction will provide information and guidance on dealing with online victimization and the associated stress.

DETAILED DESCRIPTION:
This study proposes to determine the feasibility and target engagement of a specialized chatbot intervention named SMILEY in reducing online victimization and stress among marginalized youth, including those who are Black, Hispanic, and LGBTQ+, and experiencing depression and online victimization. The primary inquiry of this study is whether SMILEY can enhance the safety and decrease stress levels in online environments for marginalized youth coping with depression and online victimization.

Pilot trial: Randomizing 2 to 1 in this study using Efron&amp;amp;amp;amp;amp;amp;amp;#39;s biased coin toss procedure. Age groups will be balanced (12-14 years old versus 15-18 years old) given that the nature of online victimization and platforms on which it occurs differ across adolescent development, racial/ethnic minority backgrounds, and sexual and gender minority backgrounds.

Sample size and power considerations: Participants (n=75; 2:1 randomization) will be identified during screening for the ETUDES Center Primary Care Study who meet inclusion criteria.

Participant groups:

A. Intervention Group: Participants will engage with SMILEY for support, in addition to receiving brief psychoeducation.

B. Control Group: Participants will only receive brief psychoeducation, without access to SMILEY

In support of the feasibility of recruitment, among patients with a PHQ-9-M scores ≥ 11 in our specialty mental health clinic for depression, 25% reported at least one OV event in the past month. Participants will be 35% Black and 10% Hispanic; given previous research, investigators expect 30% will identify as SGM. To safeguard privacy for SGM adolescents who are not out to caregivers, SGM identity will be assessed with the adolescent alone and it is not an inclusion criterion for this study. Exclusion criteria for youth are the same as for the ETUDES Center Primary Care Study, namely, mania, psychosis, developmental disability precluding comprehension of study procedures, and lack of English fluency.

Investigators anticipate that feasibility will be high (completion 50%; attrition 20%, ratings 80%); acceptability (ratings 80%); appropriateness (ratings 80%). Youth who receive SMILEY will show greater reductions in perceived stress related to OV (secondary outcome). Improvements in depression severity and risk for STB (tertiary outcomes) will be greater among youth randomized to SMILEY. Outcomes will be equitable by race and SGM identity. Exploratory (mechanistic): SMILEY will lead to decreased STB risk through improved social media self-efficacy and distress tolerance.

Intervention Delivery: Self-paced interaction with the SMILEY chatbot over 4 weeks. A research clinician will provide psychoeducation for youth and caregivers using web resources. Topics include social media self-efficacy (e.g., screen time management and positive online interactions) and guidance on how to respond to and cope with online victimization. Though usage and interactions will be self-paced, investigators expect participants will engage 2-3 times per week, for 5-10 minutes each session. Participants may receive reminders from the chatbot to engage, and if inactive for 1 week, a research assistant will assist with technical issues. Reports summarizing content may be provided to adolescents, caregivers, and providers at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents age 12-18
* Current moderate to severe depression (PHQ-9-M ≥ 11)
* Patients must screen positive for depression, PHQ-9-M score ≥ 11, and online victimization (OV). A positive screen will be OV that occurred "a few times" for at least one type of OV or "once" for at least two types of OV.

Exclusion Criteria:

* Conditions that might impair their ability to effectively deploy interventions, including current manic or psychotic episode, presence of a life-threatening medical condition requiring immediate treatment, intellectual or developmental disability precluding comprehension of study procedure
* Referring providers will be advised that adolescents must be capable of safely participating, specifically that they do not need urgent medical or psychiatric treatment.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Engagement with the chatbot | Baseline
  Engagement will be measured by the timestamps of usage of the intervention. Timestamps will be generated when there is a message from the user and a corresponding message from the chatbot.
Engagement with the chatbot | 1 month
  Engagement will be measured by the timestamps of usage of the intervention. Timestamps will be generated when there is a message from the user and a corresponding message from the chatbot.
Engagement with the chatbot | 3 months
  Engagement will be measured by the timestamps of usage of the intervention. Timestamps will be generated when there is a message from the user and a corresponding message from the chatbot.
Engagement with the chatbot | 6 months
  Engagement will be measured by the timestamps of usage of the intervention. Timestamps will be generated when there is a message from the user and a corresponding message from the chatbot.
Engagement with the chatbot | 12 months
  Engagement will be measured by the timestamps of usage of the intervention. Timestamps will be generated when there is a message from the user and a corresponding message from the chatbot.
Perceived satisfaction of the chatbot | Baseline
  Perceived satisfaction of the chatbot will be measured by the Post-Study System Usability Questionnaire (PSSUQ). Response options and scores include: "Strongly Agree (1)" to "Strongly Disagree (7)." Scores range from 1 to 7, with higher scores indicating lower levels of satisfaction and lower scores indicating higher levels satisfaction.
Perceived satisfaction of the chatbot | 1 month
  Perceived satisfaction of the chatbot will be measured by the Post-Study System Usability Questionnaire (PSSUQ). Response options and scores include: "Strongly Agree (1)" to "Strongly Disagree (7)." Scores range from 1 to 7, with higher scores indicating lower levels of satisfaction and lower scores indicating higher levels satisfaction.
Perceived satisfaction of the chatbot | 3 months
  Perceived satisfaction of the chatbot will be measured by the Post-Study System Usability Questionnaire (PSSUQ). Response options and scores include: "Strongly Agree (1)" to "Strongly Disagree (7)." Scores range from 1 to 7, with higher scores indicating lower levels of satisfaction and lower scores indicating higher levels satisfaction.
Perceived satisfaction of the chatbot | 6 months
  Perceived satisfaction of the chatbot will be measured by the Post-Study System Usability Questionnaire (PSSUQ). Response options and scores include: "Strongly Agree (1)" to "Strongly Disagree (7)." Scores range from 1 to 7, with higher scores indicating lower levels of satisfaction and lower scores indicating higher levels satisfaction.
Perceived satisfaction of the chatbot | 12 months
  Perceived satisfaction of the chatbot will be measured by the Post-Study System Usability Questionnaire (PSSUQ). Response options and scores include: "Strongly Agree (1)" to "Strongly Disagree (7)." Scores range from 1 to 7, with higher scores indicating lower levels of satisfaction and lower scores indicating higher levels satisfaction.

SECONDARY OUTCOMES:
Levels of general self-efficacy | Baseline
  Levels of general self-efficacy will be measured by the General Self-Efficacy Scale (GSE). Response options and scores include: "Not at all true (1)," "Hardly true (2)," "Moderately true," and "Exactly true (4)." Scores range from 10 to 40, with higher scores indicating higher levels of self-efficacy and lower scores indicating lower levels of self-efficacy.
Levels of general self-efficacy | 1 month
  Levels of general self-efficacy will be measured by the General Self-Efficacy Scale (GSE). Response options and scores include: "Not at all true (1)," "Hardly true (2)," "Moderately true," and "Exactly true (4)." Scores range from 10 to 40, with higher scores indicating higher levels of self-efficacy and lower scores indicating lower levels of self-efficacy.
Levels of general self-efficacy | 3 months
  Levels of general self-efficacy will be measured by the General Self-Efficacy Scale (GSE). Response options and scores include: "Not at all true (1)," "Hardly true (2)," "Moderately true," and "Exactly true (4)." Scores range from 10 to 40, with higher scores indicating higher levels of self-efficacy and lower scores indicating lower levels of self-efficacy.
Levels of general self-efficacy | 6 months
  Levels of general self-efficacy will be measured by the General Self-Efficacy Scale (GSE). Response options and scores include: "Not at all true (1)," "Hardly true (2)," "Moderately true," and "Exactly true (4)." Scores range from 10 to 40, with higher scores indicating higher levels of self-efficacy and lower scores indicating lower levels of self-efficacy.
Levels of general self-efficacy | 12 months
  Levels of general self-efficacy will be measured by the General Self-Efficacy Scale (GSE). Response options and scores include: "Not at all true (1)," "Hardly true (2)," "Moderately true," and "Exactly true (4)." Scores range from 10 to 40, with higher scores indicating higher levels of self-efficacy and lower scores indicating lower levels of self-efficacy.
Levels of distress tolerance | Baseline
  Levels of distress tolerance will be measured by the Distress Tolerance Scale (DTS). Response options and scores include: "Strongly Disagree (1)," "Mildly Disagree (2)," "Agree and Disagree Equally (3)," "Mildly Agree (4)," and "Strongly Agree (5)." Scores range from 1 to 5, with higher scores indicating higher levels of distress tolerance and lower scores indicating lower levels of distress tolerance.
Levels of distress tolerance | 1 month
  Levels of distress tolerance will be measured by the Distress Tolerance Scale (DTS). Response options and scores include: "Strongly Disagree (1)," "Mildly Disagree (2)," "Agree and Disagree Equally (3)," "Mildly Agree (4)," and "Strongly Agree (5)." Scores range from 1 to 5, with higher scores indicating higher levels of distress tolerance and lower scores indicating lower levels of distress tolerance.
Levels of distress tolerance | 3 months
  Levels of distress tolerance will be measured by the Distress Tolerance Scale (DTS). Response options and scores include: "Strongly Disagree (1)," "Mildly Disagree (2)," "Agree and Disagree Equally (3)," "Mildly Agree (4)," and "Strongly Agree (5)." Scores range from 1 to 5, with higher scores indicating higher levels of distress tolerance and lower scores indicating lower levels of distress tolerance.
Levels of distress tolerance | 6 months
  Levels of distress tolerance will be measured by the Distress Tolerance Scale (DTS). Response options and scores include: "Strongly Disagree (1)," "Mildly Disagree (2)," "Agree and Disagree Equally (3)," "Mildly Agree (4)," and "Strongly Agree (5)." Scores range from 1 to 5, with higher scores indicating higher levels of distress tolerance and lower scores indicating lower levels of distress tolerance.
Levels of distress tolerance | 12 months
  Levels of distress tolerance will be measured by the Distress Tolerance Scale (DTS). Response options and scores include: "Strongly Disagree (1)," "Mildly Disagree (2)," "Agree and Disagree Equally (3)," "Mildly Agree (4)," and "Strongly Agree (5)." Scores range from 1 to 5, with higher scores indicating higher levels of distress tolerance and lower scores indicating lower levels of distress tolerance.

OTHER OUTCOMES:
Severity of depression | Baseline
  Severity of depression will be measured by the Patient Health Questionnaire-9: Modified for Teens (PHQ-9 M). Response options and scores include: "Not at all (0)," "Several days (1)," "More than half the days (2)," and "Nearly every day (3)." Scores range from 0 to 27, with higher scores indicating higher levels of depression severity and lower scores indicating lower levels of depression severity.
Severity of depression | 1 month
  Severity of depression will be measured by the Patient Health Questionnaire-9: Modified for Teens (PHQ-9 M). Response options and scores include: "Not at all (0)," "Several days (1)," "More than half the days (2)," and "Nearly every day (3)." Scores range from 0 to 27, with higher scores indicating higher levels of depression severity and lower scores indicating lower levels of depression severity.
Severity of depression | 3 months
  Severity of depression will be measured by the Patient Health Questionnaire-9: Modified for Teens (PHQ-9 M). Response options and scores include: "Not at all (0)," "Several days (1)," "More than half the days (2)," and "Nearly every day (3)." Scores range from 0 to 27, with higher scores indicating higher levels of depression severity and lower scores indicating lower levels of depression severity.
Severity of depression | 6 months
  Severity of depression will be measured by the Patient Health Questionnaire-9: Modified for Teens (PHQ-9 M). Response options and scores include: "Not at all (0)," "Several days (1)," "More than half the days (2)," and "Nearly every day (3)." Scores range from 0 to 27, with higher scores indicating higher levels of depression severity and lower scores indicating lower levels of depression severity.
Severity of depression | 12 months
  Severity of depression will be measured by the Patient Health Questionnaire-9: Modified for Teens (PHQ-9 M). Response options and scores include: "Not at all (0)," "Several days (1)," "More than half the days (2)," and "Nearly every day (3)." Scores range from 0 to 27, with higher scores indicating higher levels of depression severity and lower scores indicating lower levels of depression severity.
Severity of suicidal ideation and behavior | Baseline
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Severity of suicidal ideation and behavior | 1 month
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Severity of suicidal ideation and behavior | 3 months
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Severity of suicidal ideation and behavior | 6 months
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.
Severity of suicidal ideation and behavior | 12 months
  Severity of suicidal ideation and behavior will be measured with the Columbia Suicide Severity Rating Scale (C-SSRS), an interviewer-rated measure. Presence of suicidal ideation and behavior will be indicated with yes/no response options. Intensity of ideation will be rated on a scale from 1-5 with higher numbers reflecting higher levels of intensity and lower numbers reflecting lower levels of intensity.

CONTACTS AND LOCATIONS:
Overall Officials: César G Escobar-Viera, MD, PhD, Principal Investigator — University of Pittsburgh; Candice Biernesser, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Western Psychiatric Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Consistent with the NIMH's data sharing and data use policies this research study and clinical trial will be compliant with requirements for depositing data with the NIMH Data Archive (NDA) in the National Database for Clinical Trials Related to Mental Illness (NDCT). Specific statements will be added to the consent forms to allow for data sharing. The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies.
Time Frame: July, 2024

DOCUMENTS (2):
  • Study Protocol (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT06835985/Prot_000.pdf
  • Informed Consent Form (2025-01-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT06835985/ICF_001.pdf